CLINICAL TRIAL: NCT02418286
Title: KLOS Study - Korean Medicine Registry for Low Back Pain Patients, a Prospective, Observational, Multicenter, Pilot Study
Acronym: KLOS
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Sangji University Oriental Medical Center, Korea (Unknown); Semyung University Korean Medicine Hospital in Chungju, Korea (Unknown); Kyunghee University Medical Center (Other); Woosuk University Oriental Medical Center, Korea (Unknown); Daejeon University (Other); Pusan National University Korean Medicine Hospital, Korea (Unknown)
Responsible Party: Principal Investigator, Yun-Kyung Song, KMD, PhD, Gachon University Gil Oriental Medical Hospital
Other Study IDs: 14-102
Record Dates: First submitted 2015-04-06; First posted 2015-04-16 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain; Back Pain; Pain; Neurologic Manifestations; Nervous System Diseases
Keywords: Low Back Pain; Korean Rehabilitation Clinic; Patient Registry
MeSH Terms: conditions — Low Back Pain; Back Pain; Pain; Neurologic Manifestations; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low Back Pain Participant Registry: Patients with low back pain in traditional Korean medicine rehabilitation clinic
  Interventions: Other: expose to any drugs or procedures based on traditional Korean medicine theory

INTERVENTIONS:
Other: expose to any drugs or procedures based on traditional Korean medicine theory — There are no specific interventions associated with this registry as it is purely observational study of medical utilization.

SUMMARY:
The Purpose of this trial is to define the characteristics of the in/outpatients with low back pain in traditional Korean medicine rehabilitation clinic. This information will create a registry that will help us to compare similarities and differences in patients and their symptoms. The more patients the investigators are able to enter into the registry, the more the investigators will be able to understand the low back pain and learn better ways of caring for patients.

DETAILED DESCRIPTION:
KLOS, prospective, multi-center, patient registry pilot study will collaborate with 7 Korean medicine hospitals and plan to recruit low back pain patients into the registry. 150 eligible patients with new episode of LBP who visit Korean medicine hospital without any other treatment history will enroll to the registry. After enrollment, study collect the individual characteristics of patient's status such as pain intensity, LBP related daily disability, anthropometrics, HRQoL at baseline, 30 and 90 days. We also access to the patient's clinical and administrative electronic records to analyze the pattern of patients' resource utilization. Overall, the aims of KLOS are to: 1) explore the general characteristics of new episode of LBP patients and; 2) evaluate the efficacy and safety of various Korean medicine treatments on low back pain based on nationwide registry outcome collecting process.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with chief complaint of low back pain in Korean medicine rehabilitation center
* Age greater than or equal to 19
* Ability to have normal communication
* Ability to give informed consent

Exclusion Criteria:

* Patients with low back pain which caused by other diseases(ex. lumbar herniated disc-surgery within past 3 months, vertebral fracture, inflammatory spondylitis, spinal infection, metastatic cancer etc.);
* Patient with musculoskeletal pain which is more severe than lower back pain;
* Patients with chronic disease may affect the results of clinical trial;
* Treated with medication for low back pain within past 4 months;
* Participated in other low back pain clinical trials within past 1 month;
* Patients who are Inability to communicate, such as alzheimer's disease or mild cognitive impairment;
* Pregnant women;
* Patients who are judged to be inappropriate for the clinical study by the researchers

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain who are visiting oriental rehabiliation clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-03; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in 'Roland Morris Disability Questionnaire' | at Baseline, 30 days after registration
  This is a self-reported questionnaire consisting of 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, bending over, sitting, lying down, dressing, sleeping, self-care and daily activities.

OTHER OUTCOMES:
Change from Baseline in 'Roland Morris Disability Questionnaire' | at Baseline, 90 days after registration
  This is a self-reported questionnaire consisting of 24 items reflecting limitations in different activities of daily living attributed to low back pain
Change from Baseline in Numeric Rating Scale of Pain | at Baseline, 30 days after registration and 90 days after registration
  A 10-point Numerical Pain Rating Scale (NRS; 0: no pain, 10: maximum pain) assesses the patients' current level of pain.
Change from Baseline in European Quality of life 5 Dimension | at Baseline, 30 days after registration and 90 days after registration
  The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Kyung Song, KMD, PhD, Professor, Principal Investigator — Gachon University, Gil Oriental Medical Center
Locations (1):
- Gachon University, Gil Oriental Medicine Center, Incheon, South Korea

REFERENCES:
- [Derived] Ko Y, Jang BH, Oh MS, Shin BC, Kim SJ, Cha YY, Ko YS, Hwang EH, Lee EJ, Jung JY, Song YK, Ko SG. Korean medicine registry for low back pain - A study protocol for prospective observational multi-center study (KLOS). Integr Med Res. 2020 Dec;9(4):100448. doi: 10.1016/j.imr.2020.100448. Epub 2020 Jun 8. PMID 32695577